CLINICAL TRIAL: NCT02337426
Title: Phase I Trial of Dimethyl Fumarate, Temozolomide, and Radiation Therapy in Glioblastoma Multiforme
Brief Title: Dimethyl Fumarate, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13-09950; NCI-2014-02619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HM20003022; MCC-13-09950 (Other: Virginia Commonwealth University/Massey Cancer Center); P30CA016059 (NIH)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Adult Brain Glioblastoma; Adult Giant Cell Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Dimethyl Fumarate; Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dimethyl fumarate, temozolomide, radiation therapy) (Experimental): CONCOMITANT THERAPY: Between 21 days (3 weeks) and 42 days (6 weeks) following the last surgical procedure, patients receive temozolomide PO QD for 42-49 days and dimethyl fumarate PO BID or TID continuously. Patients also undergo radiation therapy 5 days a week over 6 weeks for a total of 30 fractions
  MAINTENANCE THERAPY: Patients continue to receive dimethyl fumarate PO BID or TID continuously. Four weeks after completing concomitant temozolomide and radiation therapy, patients also receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dimethyl Fumarate; Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Dimethyl Fumarate — Given PO
  Other Names: Fumaric Acid, Dimethyl Ester
Drug: Temozolomide — Given PO
  Other Names: TMZ
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT

SUMMARY:
This phase 1 trial studies the side effects and best dose of dimethyl fumarate when given together with temozolomide and radiation therapy(RT) in treating patients with newly diagnosed glioblastoma multiforme (GBM). Dimethyl fumarate may help radiation therapy work better by making tumor cells more sensitive to the radiation therapy. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving dimethyl fumarate with temozolomide and radiation therapy may work better in treating glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of dimethyl fumarate (DMF) when combined with standard concurrent temozolomide and RT in subjects with newly diagnosed glioblastoma multiforme (GBM).

SECONDARY OBJECTIVES:

I. To evaluate the safety, tolerance, and toxicity of DMF when combined with standard concurrent temozolomide and RT in subjects with newly diagnosed GBM.

II. To obtain a preliminary estimate of the efficacy of DMF when combined with standard concurrent temozolomide and RT in subjects with newly diagnosed GBM.

OUTLINE: This is a dose-escalation study of dimethyl fumarate.

CONCOMITANT THERAPY: Between 21 days (3 weeks) and 42 days (6 weeks) following the last surgical procedure, patients receive temozolomide orally (PO) once daily (QD) for 42-49 days and dimethyl fumarate PO twice daily (BID) or thrice daily (TID) continuously. Patients also undergo radiation therapy 5 days a week over 6 weeks for a total of 30 fractions.

MAINTENANCE THERAPY: Patients continue to receive dimethyl fumarate PO BID or TID continuously. Four weeks after completing concomitant temozolomide and radiation therapy, patients also receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma or gliosarcoma (World Health Organization [WHO] grade IV) following either a surgical resection or biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Subjects must have recovered from surgery or biopsy before study registration
* Therapy must begin between 21 days (3 weeks) and 42 days (6 weeks) after the most recent brain tumor surgery(resection or biopsy)
* Documentation of steroid doses 10-14 days prior to study registration and stable or decreasing steroid dose over the week prior to registration
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3 (untransfused)
* Hemoglobin >= 10 g/dL (the use of transfusion or other intervention to achieve hemoglobin >= 10 g/dL is acceptable)
* Creatinine =< 1.5 x upper limit of normal (ULN) for the laboratory or calculated or actual creatinine clearance > 45 mL/min
* Total bilirubin =< 1.5 x ULN for the laboratory (total bilirubin criteria may be waived if a subject has documented Gilbert's syndrome)
* Aspartate aminotransferase (AST) =< 3 x ULN for the laboratory
* Alanine aminotransferase (ALT) =< 3 x ULN for the laboratory
* Women of childbearing potential and male subjects must practice adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanoma skin cancer) unless disease free for >= 3 years
* Recurrent malignant gliomas
* Metastases detected below the tentorium or beyond the cranial vault
* Prior chemotherapy or radiation therapy (RT) for the diagnosis of GBM or for cancers of the head and neck
* Clinically significant cardiac disease, including major cardiac dysfunction, such as uncontrolled angina, clinical congestive heart failure with New York Heart Association (NYHA) class III or IV, ventricular arrhythmias requiring anti-arrhythmic therapy
* Pregnant or lactating women
* History of allergic reactions or intolerance to any of the required agents on the study
* History of hypersensitivity to dacarbazine
* Any treatment for GBM, other than surgery or anti-epileptic therapy, within 30 days prior to study treatment initiation
* Other condition(s) that in the opinion of the investigator might compromise the objectives of the study or increase patient risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
RP2D for DMF when combined with concurrent temozolomide and radiotherapy determined by the incidence of dose limiting toxicities (DLTs) graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to 6 weeks
  Subjects' treatment dosing level, dose modification, DLTs, and evaluability for DLTs and response will be listed and summarized by basic descriptive statistics (such as frequency and proportion).

SECONDARY OUTCOMES:
Incidence of adverse events graded according to NCI CTCAE version 4.0 | Up to 30 days after completion of treatment
  Subjects' demographics, adverse events, serious adverse events, and treatment status will be listed and summarized by descriptive statistics (such as frequency, proportion, mean, standard deviation, median, and range).
Progression free survival (PFS) | Time from registration to time of symptomatic and/or radiographic progression or death, whichever occurs first, assessed up to 2 years
  The Kaplan-Meier method will be conducted to describe PFS, and median PFS will be estimated, along with 95% confidence intervals. A Cox regression model may be used to model the PFS and adjusting for any effects of potential clinical characteristics.
Overall survival (OS) | Time from registration until death from any cause, assessed up to 2 years
  The Kaplan-Meier method will be conducted to describe OS, and median OS will be estimated, along with 95% confidence intervals. A Cox regression model may be used to model the OS and adjusting for any effects of potential clinical characteristics.
Response rate assessed as per the Response Assessment in Neuro-oncology for magnetic resonance imaging scans or Macdonald criteria for computed tomography scans | Up to 2 years
  The clinical response rate will be calculated for each cohort, along with their corresponding 95% confidence intervals. Logistic regression may be used to model the rate by adjusting potential clinical characteristics (such as age, gender, and tumor grade). Mean and standard deviation of duration of response (overall response, complete response, and stable disease, respectively), along with its 95% confidence interval, will be estimated based on the method proposed by Ellis et al. via the exponential distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Malkin, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States